CLINICAL TRIAL: NCT06790056
Title: Efficacy of Endoscopic Band Ligation (DEBL) for Duodenal Neuroendocrine Neoplasms(dNENs) : A Prospective Study
Brief Title: Efficacy of Endoscopic Band Ligation (DEBL) for Duodenal Neuroendocrine Neoplasms(dNENs)
Acronym: DEBL
Status: Completed | Type: Observational
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Mohan Ramchandani, Consultant Gastroenterologist, Asian Institute of Gastroenterology, India
Other Study IDs: DEBL- 01
Record Dates: First submitted 2024-01-11; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Duodenal Neuroendocrine Tumor
Keywords: lesion size,; tumour; binding
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Duodenal endoscopic band ligation group: We will collect your basic demographics details like age, Sex, date of admission, Endoscopy (is a test to look inside your body) details of Site, size, number of lesion.
  By EUS (Endoscopic ultrasound (EUS) combines two techniques - endoscopy and ultrasound - to help doctors see, evaluate and diagnose conditions in and near the gastrointestinal (GI) tract) details of layer of Duodenum involved, site/size/number of lesions.
  We will collect your details of Duodenal endoscopic band ligation procedure to check feasibility, technical success.
  You are requested to come for follow up for 3 months for endoscopy prodecure.
  Interventions: Procedure: duodenal ndoscopic bind ligation

INTERVENTIONS:
Procedure: duodenal ndoscopic bind ligation — We will collect your basic demographics details like age, Sex, date of admission, Endoscopy (is a test to look inside your body) details of Site, size, number of lesion.
  By EUS (Endoscopic ultrasound (EUS) combines two techniques - endoscopy and ultrasound - to help doctors see, evaluate and diagnose conditions in and near the gastrointestinal (GI) tract) details of layer of Duodenum involved, site/size/number of lesions.
  We will collect your details of Duodenal endoscopic band ligation procedure to check feasibility, technical success.
  You are requested to come for follow up for 3 months for endoscopy prodecure.

SUMMARY:
Primary objective To evaluate the therapeutic efficacy (clinical success) of dEBL at 3 months

2b. Secondary objective

To evaluate adverse events, technical success and recurrence on follow-up

50 patients over 1-year duration based on our previous study of Prospective data (2023-2024)

DETAILED DESCRIPTION:
We will collect your basic demographics details like age, Sex, date of admission, Endoscopy (is a test to look inside your body) details of Site, size, number of lesion.

By EUS (Endoscopic ultrasound (EUS) combines two techniques - endoscopy and ultrasound - to help doctors see, evaluate and diagnose conditions in and near the gastrointestinal (GI) tract) details of layer of Duodenum involved, site/size/number of lesions.

We will collect your details of Duodenal endoscopic band ligation procedure to check feasibility, technical success.

You are requested to come for follow up for 3 months for endoscopy prodecure.

ELIGIBILITY:
Inclusion Criteria:

* Patients age >18 years
* Size of lesion less than 15mm
* Site of lesion- duodenum (d1-d4)
* No of lesions- ≤6

Exclusion Criteria:

* Age less than 18 years
* Non-duodenal lesion
* Local or distant metastasis
* Lumen occluding lesions
* Uncorrectable coagulopathy
* Not willing for consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 50 patients over 1-year duration .
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-02-29 (Actual); Primary Completion 2024-11-10 (Actual); Study Completion 2024-11-11 (Actual)

PRIMARY OUTCOMES:
Therapeutic efficacy (clinical success) of dEBL at 3 months and 1 year | One year
  Therapeutic efficacy (clinical success) of dEBL at 3 months and 1 year

SECONDARY OUTCOMES:
Adverse events and recurrence on follow up | One year
  Univariate and multivariate analysis will be done to determine which are the factors associated with clinical success and clinical recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Hardik Rughwani, Principal Investigator — AIG HOSPITALS
Locations (1):
- Hardik Rughwani, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No